CLINICAL TRIAL: NCT06028009
Title: Vaginal Injection of Platelet Rich Plasma (PRP) for the Genitourinary Syndrome of Menopause (GSM)
Brief Title: PRP Injections for Genitourinary Syndrome of Menopause
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006805
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: PRP; Sexual Function Disturbances; Genitourinary Syndrome of Menopause; Postmenopausal Symptoms; Vaginal Atrophy
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich plasma injection (Experimental)
  Interventions: Procedure: Injection of platelet-rich plasma
- 0.9% saline injection (Sham Comparator)
  Interventions: Procedure: Injection of saline

INTERVENTIONS:
Procedure: Injection of platelet-rich plasma — Injection of autologous platelet-rich plasma into anterior vaginal wall
  Arms: Platelet-rich plasma injection
Procedure: Injection of saline — Injection of sterile normal saline into anterior vaginal wall
  Arms: 0.9% saline injection

SUMMARY:
Platelet-rich plasma (PRP) is autologous blood which has been centrifuged to separate the supernatant resulting in a solution with high concentration of platelets. Injection of PRP stimulates cell growth and can has been proven safe and effective for uses in orthopedics, dermatology, and gynecology. Despite the relative paucity of data, the use of PRP as a therapy for sexual dysfunction and genitourinary symptoms in the setting of menopause has been patented as the O-Shot and V-Shot. This is a single-blinded randomized control trial to determine if PRP injections into the anterior vaginal wall improve sexual functioning in women diagnosed with the genitourinary syndrome of menopause (GSM) characterized by vaginal dryness/irritation.

ELIGIBILITY:
Inclusion Criteria:

* Women (assigned female at birth) at least 18 years old with a clinical diagnosis of GSM
* Sexually active with at least one episode of sexual activity per week in the preceding 4 weeks defined as follows: Partnered or solo penetrative or non-penetrative stimulation of the clitoris or vagina
* English-speaking
* Willingness and able to comply with the study requirements

Exclusion Criteria:

* Symptomatic pelvic organ prolapse protruding beyond the hymen)
* History of prior vaginal mesh or midurethral mesh sling surgery
* History of pelvic radiation or genital tract malignancy
* Current symptomatic pelvic organ prolapse (stage II or greater)
* Active vulvar dermatoses or genitourinary infection
* Unable to hold anticoagulation
* Hormonal replacement therapy (systemic, local, or vaginal) within 3 months of participation
* Pregnancy or pre-menopausal status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | Assessed at baseline and at 6 weeks and 6 months post-procedure
  Validated questionnaire to assess domains of sexual function with range from 2 to 36 with lower score indicating worse sexual functioning (diagnostic for sexual dysfunction if score is less than or equal to 26.55)

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | Assessed at 6 weeks and 6 months post-intervention
  Single item questionnaire evaluating improvement in vaginal dryness with scale from 1 to 7 with lower score indicating greater improvement in vaginal dryness
Visual analog scale for vaginal dryness (VAS) | Assessed at 6 weeks and 6 months post-intervention
  Visual analog scale for vaginal dryness (VAS) with range from 0 to 10 with higher score indicating higher degree of bothersome vaginal dryness
Urinary Distress Inventory (short form) (UDI-6) | Assessed at baseline and 6 weeks/6 months post-intervention
  6 item questionnaire assessing urinary symptoms with range from 0-18 with higher score indicating greater distress related to urinary symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Lafayette Medical Centre, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No